CLINICAL TRIAL: NCT00665886
Title: Randomized Study of Closed Peripheral Intravenous Systems Versus Mounted Open Systems
Brief Title: Compact Closed System Versus Mounted Open System (COSMOS)
Acronym: COSMOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Foundation for Biomedical Research and Innovation (Other)
Responsible Party: Juan Luís González López/Materials Resources Coordinator, Hospital Clínico San Carlos de Madrid (Spain)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HCSC-DIRENF-0802; P-08/014
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2009-04-13 (Estimated); Status verified 2009-04

CONDITIONS: Catheterization, Peripheral
Keywords: Peripheral venous catheter; Catheter-related complication; Bacterial Colonization; Dwell time; Closed system; Costs; Polyurethane; Teflon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Experimental Group (Closed System):
  Nexiva® Safety IV Catheter from BD (Becton Dickinson). The catheter has wings, a passive safety feature, an integrated Y extension tubing integrated and needle-less access using a split septum BD QSyte®. In order to completely close the Y connector a second Q-Syte® is added from the moment of catheter insertion
  Interventions: Device: Closed Intravenous System - Nexiva®
- 2 (Active Comparator): Control group (Open System):
  A 'mounted' system consisting of the Vasocan® Safety catheter of B. Braun Medical, SA. To the control catheters a three-way tap ('stopcock') with extension tubing 10 cm long (Connecta® Extra 3, from BD) is added. This comes as one unit (tap and tubing are integrated). When not in use the three-way tap ('stopcock') remains closed using a red cork Luer/Luer-Lock Sollner®, made by Amebil, SA.
  Interventions: Device: Open Intravenous System - Vasocan®

INTERVENTIONS:
Device: Open Intravenous System - Vasocan® — Vasocan® Safety catheter 18 G x 45 mm (Ref. 4248139S), 20 G x 33 mm (Ref. 4248112S) y 22 G x 25 mm (Ref. 4248090S)with wings and a passive safety mechanism. To the control catheters a three-way tap ('stopcock') with extension tubing 10 cm long (Connecta® Extra 3) from BD (ref 394995)will be added.
  Other Names: Vasocan® Safety catheter of B. Braun Medical; Connecta® Extra 3 of BD; Luer/Luer-Lock of Sollner®
  Arms: 2
Device: Closed Intravenous System - Nexiva® — BD Nexiva® Catheter (18G x 45 mm, 20 G x 32 mm, 22 G x 25 mm) (Ref. 383609,Ref. 383606,Ref. 383602) BD QSyte®, Ref. 385100 Catheter material is Vialon®. The entire system is Latex and PVC free.
  Other Names: Nexiva®; QSyte®.
  Arms: 1

SUMMARY:
The purpose of this study is to investigate, in a prospective and randomized fashion, the clinical performance of a closed intravenous system versus an open conventional one, with respect to ease of handling and effectiveness (as defined by time of survival without complications), security provided to professionals and patients against accidental blood exposure or needlestick injury, catheter-related complications such as phlebitis, pain and blockage and overall costs of the two systems.

DETAILED DESCRIPTION:
Study Design:

This study has a prospective, open, randomized, unblinded, group-sequential design. Study initiation will be proceeded by a program of education and training for all the nurse participants to ensure proper handling of both systems and standard insertion and maintenance techniques for both catheter systems. This standardization will include disinfection of the skin and access ports as well as fixation of the catheter using a standard transparent dressing. Also training will be given on best practice procedures for removing the catheter, on sterile technique for culture of the catheter tip and on proper data capture methods using the Clinical Report Form (CRF). All the nurses participating in the study will certify their attendance to all trainings, their acceptance of the present protocol and their voluntary participation by signing the Participant Registry at the conclusion of the trainings. They must give their full names as well as personnel and unit numbers, which will then be used to constitute the Investigating Group as well as to protect identities while providing a traceable record of participants.They must have passed a training examination consisting of 10 questions related to the study with a passing mark of at least 80% questions correct. The study will be preformed in three medical and surgical units of the University Clinical Hospital San Carlos of Madrid, which is affiliated with the Madrid Health Service, and is an integral part of the Autonomous Region (Community) of Madrid.Trainings and other activities related to the study will not begin until formal approval of the protocol by the Ethics Committee (abbreviated CEIC in Spanish) of this hospital. In order to reduce variability in the study, all catheters will be inserted using only 70% alcohol for disinfection of the skin and access ports.

Following manufacturer recommendations, all three-way taps (in USA, 'stop cocks') with extension tubes will be changed every 72 hours and split-septum connectors will be changed every 8 days. In order to calculate colonization rates in both catheter systems and the correlation of colonization with clinical complications, tip cultures will be taken of a representative sample of catheters in each arm. This process will be randomized and will coincide with catheter withdrawal. Additionally all catheters removed because of pain, phlebitis or suspected infection will have their tips cultured. Our sample size target for cultured tips is 380 in total. During the study, six nurse-coordinators, with experience in intravenous therapy and special training in study procedures, will actively supervise all aspects of catheter management and will report to the Principal Investigator (PI) on a regular basis. They will ensure the randomization processes are followed and that all procedures established by the Protocol, as well as of the correct filling out of the CRF, are rigorously adhered to. In order to accomplish this they will make daily inspections of all catheters included in the study, will check each item on each CRF daily to ensure all are properly and promptly filled out and will follow the catheter tip cultures to certify that the results are registered on the CRFs. The coordinators will not otherwise intervene in patient care. Any decision related to placing or removing a peripheral catheter for any cause, all decisions on the care and maintenance of the catheter system, and all treatment decisions related to the patients will be the sole responsibility of the doctors and nurses caring for the patient. Nurse-coordinators and/or the PI will not intrude in any way in these decisions. An intermediate analysis will be done when each unit reaches 166 catheters inserted. This analysis will allow us to confirm the power calculation of the study and determine final sample size targets. All patients admitted to one of the three participating units, who needs a peripheral venous catheter of gauge size18 G, 20 G or 22 G, will be evaluated for potential inclusion in the study. Using the CRF a determination of eligibility will be made and then study purpose and requirements will be explained in layman's terms to the patient by his primary nurse. If accepted into the study patient informed consent will be obtained. Informed consent may be verbal on the condition that it is witnessed by one of his or her relatives and is documented in the CRF. After this the patient will be randomized to the experimental group (closed system) or to the control (open system).

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to one of the participating units: H2N (Internal Medicine), H3N (Urology, Surgery, Trauma) and H3S (General Surgery)
* Age equal to or greater than 18 years
* Clinical need for a peripheral catheter of gauge size 18 G to 22 G for an anticipated period of 24 hours or greater
* Informed verbal consent before a witness (family relative or a health care professional employed by the hospital)

Exclusion Criteria:

* Minor (<18 years old)
* Inability to understand the information regarding study purpose and procedure
* Absence of witnessed verbal informed consent
* Participation in any other study
* IV placed under emergency conditions
* Presence of a Central Venous Catheter or PICC line
* Presence of a fever of 38º C of more at the time of inclusion
* Anticipated use of the catheter and/or stay in the unit of less than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Length of time catheter remains in place without clinical symptoms | For the individual patient: Dwell time of the catheter free of complications, defined as the average time in hours from the insertion to the withdrawal of the catheter. For the study itself: From March through June, 2008.

SECONDARY OUTCOMES:
Incidence of complications of the catheter, bacterial colonization of catheter tips and costs of therapy. | For an individual patient: From the randomized insertion of the catheter until its withdrawal. For the study itself: From March through June, 2008.

CONTACTS AND LOCATIONS:
Overall Officials: Juan L Gonzalez Lopez, M.A. Nurse, Study Chair — Hospital Clínico San Carlos (Madrid, Spain); Juan Luis González López, M.A. Nurse, Principal Investigator — Hospital Clínico San Carlos (Madrid, Spain)
Locations (1):
- Hospital Clínico San Carlos, Madrid, Madrid, Spain